CLINICAL TRIAL: NCT07109245
Title: Do Antipsychotics Block Insulin Action in the Brain: is it a Class Effect?
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 2025/010
Record Dates: First submitted 2025-07-17; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Brain Insulin Sensitivity; Healthy Controls; Cognition
Keywords: Brain Insulin Sensitivity; Healthy Control Study; Haloperidol; Cognition; MRI
MeSH Terms: interventions — Haloperidol; Insulin Lispro; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Haloperidol (Experimental): The oral investigational agent haloperidol (Generic Brand: TEVA-HALOPERIDOL) will be self-administered, at night, over 7 days. Haloperidol will be titrated up to 2 mg.
  Interventions: Drug: Haloperidol; Drug: Insulin Lispro; Other: Saline
- Placebo (Placebo Comparator): Placebo capsules, visually identical to those containing haloperidol, will be administered according to the same dosing schedule
  Interventions: Drug: Placebo; Drug: Insulin Lispro; Other: Saline

INTERVENTIONS:
Drug: Haloperidol — The oral investigational agent haloperidol (Generic Brand: TEVA-HALOPERIDOL) will be self-administered, at night, over 7 days. Haloperidol will be titrated up to 2 mg.
  Arms: Haloperidol
Drug: Placebo — Oral placebo, encapsulated and to be taken at an equivalent titration schedule to Haloperidol.
  Arms: Placebo
Drug: Insulin Lispro — A total of 160 IU of intransal insulin (=1.6 mL) will be administered on MRI scanning visits (80 IU = 0.8 mL delivered per nostril). Humalog; Eli Lilly Canada
Other: Saline — A total of 1.6 mL of intranasal saline will be administered on each MRI scanning visit (0.8 mL delivered per nostril).

SUMMARY:
This study aimed at helping researchers understand how a medication called haloperidol can affect insulin action in the brain. Insulin is a hormone in the body that controls sugar levels in part by lowering the amount of glucose produced by the liver. After eating a meal, insulin levels go up in both the blood and the brain. Insulin in the brain has also been shown to affect the way the brain works and processes information (also known as "cognition"). Haloperidol, is an antipsychotic medication used to treat a variety of disorders such as schizophrenia spectrum disorders, bipolar disorder, and major depressive disorder, but long-term use can have metabolic side effects, like weight gain, type 2 diabetes, and cardiovascular disease. The purpose of this study is to investigate how antipsychotic medications, such as haloperidol, which carries the risk of metabolic changes, might interrupt the effect of insulin action in the brain. This will help researchers learn how to potentially reduce metabolic risk for people who take these kinds of medications in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Must be deemed to have the capacity to provide informed consent
2. Must sign and date the informed consent form
3. Stated willingness to comply with all study procedures;
4. Age: 18-35
5. Body Mass Index (BMI) 18.5-24.9 kg/m2
6. Both sexes

Exclusion Criteria:

1. History of psychiatric illness, including any substance use (screened using the Mini International Neuropsychiatric Interview (MINI))
2. Pre-diabetes or diabetes (fasting glucose ≥6.0 mmol/L, HbA1c>6% or use of anti-diabetic drug),
3. Evidence of impaired insulin sensitivity, assessed using the Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) ≥2.5
4. Family history of diabetes in a first degree relative (parent or sibling)
5. Use of weight reducing agents
6. History of kidney or liver disease
7. History of cell blood disorders
8. Irregular menstrual cycles (e.g., menstruation occurs less than 21 days or more than 35 days apart, or not having menstruated for three months (or 90 days), or conditions such as endometriosis or polycystic ovary syndrome (PCOS) or prior surgical interventions such as a hysterectomy or oophorectomy)
9. Current use of hormonal birth control (e.g., pill, patch, hormonal intrauterine device [IUD], ring). Participants must have had at least 2 regular menstrual cycles following the discontinuation of hormonal birth control [50]
10. Current use of progesterone, estrogen, testosterone, or fertility treatment.
11. Pregnant, gave birth in the last year, or breastfeeding. Participants must have at least 3 regular menstrual cycles post-breastfeeding before beginning the study.
12. Major medical or surgical event within the last 6 months
13. Contraindications for MRI, including metal implants, pacemakers, cochlear implants, claustrophobia, weight >250 lbs
14. Any contraindications to the investigational products as listed in the product monographs including known hypersensitivity to the drug or the excipients of the product (note: enzymatic lactose intolerance is NOT exclusionary),
15. Any medications that increases risk of hypoglycemia or could contribute to hyperglycemia
16. Any medical conditions that constitute as a warning/precaution for haloperidol, lorazepam, benztropine, or insulin.
17. Use of any of the prohibited medications listed in the product monograph of haloperidol, lorazepam, benztropine, or insulin (Pheochromocytoma, barbiturates, and narcotics are exclusionary, any use of painkillers and antihistamines must be reviewed by PI but are not exclusionary

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
RsFC between the anterior cingulate cortex of the salience network and the lateral parietal cortex of the DMN | From enrollment to the end of study will be up to 5 months
  Resting state functional connectivity (rsFC) between the anterior cingulate cortex of the salience network and the lateral parietal cortex of the default mode network (DMN) will be assessed through a MRI-based assay. Calculated using the correlation between two brain regions' blood-oxygen-level-dependent (BOLD) signal times.
Metabolic Outcome: BMI | From enrollment to the end of study will be up to 5 months
  Weight (kg) and Height (cm) will be aggregated to BMI (kg/m^2) at screening and MRI scanning visits.
Metabolic Outcome: Waist Circumference | From enrollment to the end of study will be up to 5 months
  Waist Circumference (cm) collected at screening and MRI scanning visits.
Metabolic Outcome: Glucose | From enrollment to the end of study will be up to 5 months
  Glucose (mmol/L), will be measured at 2 time points on each MRI scanning day, pre- and post-intranasal insulin challenge.
Metabolic Outcome: Insulin | From enrollment to the end of study will be up to 5 months
  Insulin (uIU/mL), will be measured at screening and at 2 time points on each MRI scanning day, pre- and post-intranasal insulin challenge.
Metabolic Outcome: C-peptide | From enrollment to the end of study will be up to 5 months
  C-peptide (nmol/L), will be measured at screening and 2 time points on each MRI scanning day, pre- and post-intranasal insulin challenge.
Metabolic Outcome: HbA1c | From enrollment to the end of study will be up to 5 months
  HbA1c (mmol/mol), will be measured at screening and 2 time points on each MRI scanning day, pre- and post-intranasal insulin challenge
Metabolic Outcome: HOMA-IR (Homeostatic Model Assessment for Insulin Resistance) | From enrollment to the end of study will be up to 5 months
  HOMA-IR, will be measured at 2 time points on each MRI scanning day, pre- and post-intranasal insulin challenge. HOMA-IR = (Fasting Insulin (uIU/mL) * Fasting Glucose (mmol/L)) / 22.5

SECONDARY OUTCOMES:
Antipsychotic Related Outcome: Plasma antipsychotic (haloperidol) level | From enrollment to the end of study will be up to 5 months
  Plasma antipsychotic (haloperidol) levels will be measured with concentrations expressed in nanograms per millilitre (ng/mL). Collected on each MRI scanning day.
Antipsychotic Related Outcome: Stanford Sleepiness Scale | From enrollment to the end of study will be up to 5 months
  The Stanford Sleepiness Scale (SSS), which is a self-reported scale (scale of 1-7), where higher scores indicate greater sedation. Administered on each MRI scanning visit.
Antipsychotic Related Outcome: Digit Symbol Substitution Test | From enrollment to the end of study will be up to 5 months
  The Digit Symbol Substitution Test (DSST), which will be reported as the number of correct responses (count per 90 seconds), where lower scores reflect greater sedation or cognitive slowing. Administered on each MRI scanning day.
Antipsychotic Related Outcome: Barnes Akathisia Scale | From enrollment to the end of study will be up to 5 months
  The Barnes Akathisia Scale (BAS) (scale of 0-14), with higher scores indicating more severe akathisia. Administered on each MRI scanning day.
Antipsychotic Related Outcome: Simpson-Angus Scale | From enrollment to the end of study will be up to 5 months
  The Simpson-Angus Scale (SAS) (scale of 0-40), where higher values indicate more pronounced parkinsonian symptoms. Administered on each MRI scanning day.
Antipsychotic Related Outcome: Abnormal Involuntary Movement Scale | From enrollment to the end of study will be up to 5 months
  Abnormal Involuntary Movement Scale (AIMS) (scale of 0-42), with higher scores corresponding to more severe involuntary movements. Administered on each MRI scanning day.
Antipsychotic Related Outcome: UKU Side Effect Rating Scale | From enrollment to the end of study will be up to 5 months
  Side effects will be assessed using the UKU Side Effect Rating Scale, which will be reported as a scale score (scale of 0-144), where higher scores indicate a greater burden of side effects. Administered on each MRI scanning day.

CONTACTS AND LOCATIONS:
Overall Officials: Mahavir Agarwal, MBBS, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided